CLINICAL TRIAL: NCT03598556
Title: Strategies for the Prevention of Bone Loss Among Patients With HIV on Antiretroviral Therapy in China
Brief Title: Preventing Bone Loss Among Chinese Patients With HIV on ART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing YouAn Hospital (Other); Beijing Ditan Hospital (Other); Guangxi Autonomous Region Longtan Hospital (Unknown); Fuzhou Infectious Diseases Hospital (Unknown); Shenzhen Third People's Hospital (Other); Yale University (Other)
Responsible Party: Principal Investigator, LI Taisheng, Professor, Department of Infectious Diseases, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CACT 1807
Record Dates: First submitted 2018-07-15; First posted 2018-07-26 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: HIV/AIDS; Osteoporosis; Bone Loss
Keywords: China; Anti-retroviral Therapy; Vitamin D; Tenofovir; Efavirenz; Lamivudine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Osteoporosis; Bone Diseases, Metabolic | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 Supplementation Arm (Experimental): This arm will receive 180,000IU vitamin D3 every 3 months from baseline through week 96.
  Interventions: Dietary Supplement: Vitamin D3
- Placebo Arm (Placebo Comparator): This arm will receive placebo every 3 months from baseline through week 48, followed by 180,000IU vitamin D3 every 3 months from week 48 through week 96.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 180,000IU Vitamin D3 oral emulsion
  Arms: Vitamin D3 Supplementation Arm
Other: Placebo — Placebo
  Arms: Placebo Arm

SUMMARY:
The major goal of this study will be to conduct a randomized, double-blind, placebo-controlled, clinical trial of intermittent high-dose vitamin D3 supplementation (180,000IU) given at the point of care (every 3 months) after initiation of ART with tenofovir/ lamivudine/ efavirenz to compare its ability to mitigate reductions in bone mineral density over 12 months compared to placebo.

DETAILED DESCRIPTION:
Studies among adult and pediatric populations have suggested vitamin D supplementation may be efficacious for mitigating the bone loss seen with tenofovir-based antiretroviral therapy (ART). Because patients with HIV face significant pill burden, competing priorities and health care associated costs, we seek to explore a pragmatic approach to prevention. The investigators propose a randomized controlled, double-blind, placebo intervention trial to assess the efficacy, tolerability, and safety of an intermittent high-dose vitamin D3 supplementation regimen given quarterly at the point of care for adult patients receiving free ART through the China National Free AIDS Treatment Program. The period of supplementation will be limited to the first 48 weeks after treatment initiation when ART-associated bone loss is most pronounced. This will be followed by supplementation of all participants with vitamin D3 from 48 to 96 weeks to compare the impact of early vitamin D3 supplementation (at ART initiation) versus late vitamin D3 supplementation (at 48 weeks) on change in BMD.

Furthermore, despite the rapid rise in access to ART in China, infrastructure to diagnose and manage osteoporosis is not always easily accessible for patients with HIV in China due to limited availability of dual-energy x-ray absorptiometry (DXA), the gold standard for BMD measurement. Therefore, the current proposal also seeks to bridge this gap by exploring the potential applications of quantitative ultrasound (QUS), a portable and low-cost method of assessing BMD that has been demonstrated to reliably predict fracture, in HIV care settings.

A total of 400 treatment-naïve Chinese adults diagnosed with HIV from 3 study sites in Beijing will be enrolled and followed with serial DXA exams to evaluate the primary aim. These 400 patients plus another 200 participants from 3 additional study sites from Fuzhou, Shenzhen, and Guangxi province, will be evaluated with serial QUS ultrasound examinations for the secondary aims. Serum and urine samples will be collected and stored at pre-specified time points.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Willingness and availability to engage in study activities for the duration of the study
* Documented HIV-1 infection (confirmed by Western blot)
* ART naïve at the time of enrollment
* Eligible to initiate ART (TDF/3TC/EFV) within 1 month
* Ability to take oral medication and be willing to adhere to the mediation regimen
* For females of reproductive potential: use of highly effective contraception

Exclusion Criteria:

* Pregnancy or breastfeeding
* AIDS-defining illness within 2 weeks of entry
* Liver disease (transaminase and alkaline phosphatase levels more than three times the upper limit of the normal range (ULN), bilirubin level more than 2.5 times the ULN)
* Chronic kidney disease (serum creatinine level more than 1.5 times the ULN)
* Patients with a history of injection drug usage
* Known history of osteoporosis, osteoporotic fracture, or other metabolic/inherited bone disorder
* History of treatment with prescription therapies for osteoporosis (for example: bisphosphonates, denosumab, teriparatide, selective estrogen receptor modifying agents, active forms of vitamin D).
* Unwillingness to discontinue previous vitamin D supplementation, if any, at time of enrollment
* Rheumatoid arthritis
* Malabsorption or inflammatory bowel disease
* Hyperparathyroidism, hypercalcemia, or hypocalcemia
* History of kidney stones
* Poorly controlled thyroid disease
* History of neuromuscular disorder/movement disorder, stroke or seizures
* History of significant neurocognitive disorders (including mental health conditions or dementia)
* Glucocorticoids, estrogen, testosterone, or anticonvulsant use within the past six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in Bone Mineral Density (BMD) | Baseline to week 48
  In the three sites in Beijing (N=400), compare percent change in BMD at the lumbar spine and total hip, as measured by dual-energy x-ray absorptiometry (DXA) at week 48.

SECONDARY OUTCOMES:
Immediate vs. Delayed Vitamin D3 Supplementation | Weeks 48 to 96
  In the three sites in Beijing (N=400), from 48 to 96 weeks, switch the placebo arm to vitamin D3 supplementation to compare percent change in BMD at 96 weeks between patients who initiated vitamin D3 supplementation at the start of ART versus those who initiated vitamin D3 after 1 year of ART.
Change in Quantitative Ultrasound (QUS) Measures | Baseline to 96 weeks
  In all six study sites (N=600), evaluate percent change in SOS and BUA over 48 weeks in the vitamin D treatment group compared with placebo, as measured by QUS. Further, evaluate the ability of QUS to independently identify the same group of patients at greatest risk for severe bone loss, as compared with risk stratification using DXA.
Change in Biochemical Markers | Baseline to 96 weeks
  To measure the effect of the proposed intervention on markers of vitamin D and bone metabolism, inflammation and HIV disease status.

CONTACTS AND LOCATIONS:
Overall Officials: Taisheng Li, MD, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (6):
- China (6):
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fuzhou Infectious Diseases Hospital, Fuzhou, Fujian
  - Shenzhen Third Hospital, Shenzhen, Guangdong
  - Longtan Hospital, Liuchow, Guangxi Autonomous Region